CLINICAL TRIAL: NCT06308796
Title: Prevention of Caries in Head and Neck Cancer Survivors Who Underwent Radiotherapy: a Randomized Controlled Trial
Brief Title: Prevention of Caries in Head and Neck Cancer Survivors Who Underwent Radiotherapy
Acronym: RADIOCARIES
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Milan (Other)
Responsible Party: Principal Investigator, Elena Varoni, Associate Professor, University of Milan
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: RADIOCARIES2023
Record Dates: First submitted 2024-02-02; First posted 2024-03-13 (Actual); Last update posted 2024-03-15 (Actual); Status verified 2024-03

CONDITIONS: Caries,Dental; Head and Neck Cancer; Radiotherapy; Complications
MeSH Terms: conditions — Dental Caries; Head and Neck Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CaP + Fluoride (Experimental): Irradiated head and neck cancer patients receiving topical CaP mousse to be applied at home (once a day for the first 3 months, then once a day for one week per month as maintenance), besides topical fluoride (F) in form of professional varnishes (every 6 months) and home products (once a day oral rinse with F mouthwash; three times a day toothpaste with brushing).
  Interventions: Other: Application of CaP dental mousse
- Only fluoride (No Intervention): Irradiated head and neck cancer patients receiving only topical fluoride (F) in form of professional varnishes (every 6 months) and home products (once a day oral rinse with F mouthwash; three times a day toothpaste with brushing). Topical fluoride is included in the standard of care, according to national and international guidelines.

INTERVENTIONS:
Other: Application of CaP dental mousse — Application of calcium phosphate (CaP) mousse on dental surfaces at home, once a day for 3 months; followed, as maintenance, once a day for just one week a month.
  Arms: CaP + Fluoride

SUMMARY:
One of the long-term side effects of head and neck radiotherapy (RT) is radiation-induced tooth decay. Hyposalivation, associated with radiation therapy, further increases caries susceptibility and caries progression, due to the lack of salivary protective effects and of tooth minerals useful for remineralization processes, especially calcium phosphate (CaP). Dental extractions that could be required in case of severe tooth decay expose the patient to the risk of osteoradionecrosis of the jaws (i.e. the necrosis of the bone tissue following a local trauma, including surgical trauma). This protocol aims at verifying the effectiveness of CaP mousse in the prevention of carious lesions, added to topical fluoride. A randomized controlled clinical trial will be performed comparing CaP + fluoride treatment versus no treatment in head and neck cancer patients, who received radiotherapy. The hypothesis is that CaP, which is lacking in the mouth of these patients due to hyposalivation, can combine with fluoride to promote remineralization, reducing the risk of carious lesions.

ELIGIBILITY:
Inclusion Criteria:

* previous head and neck radiotherapy for oncological treatment

Exclusion Criteria:

* complete edentulism
* pregnancy or breastfeeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2023-04-01 (Actual); Primary Completion 2026-01-31 (Estimated); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
Number of new cavitated caries per each patient (incidence of caries) | Assessment every 3 months up to 2 years
  Identification of new carious lesion using International Caries Detection and Assessment System from score 0 initial lesions to 6 large cavitated lesions (ICDAS; 4-6)

SECONDARY OUTCOMES:
Number of extracted teeth per patient (incidence of extracted teeth) | Assessment every 3 months up to 2 years
  Number of new teeth extracted
Number of patients with a diagnosis of osteoradionecrosis (incidence of osteoradionecrosis) | Assessment every 3 months up to 2 years
  Number of new areas of bone necrosis
Number of dental surfaces with caries or filling, and missed teeth | Assessment every 3 months up to 2 years
  Recording of the diseased, missed, filled surfaces (DMFS) index
Rate of dentinal hypersensitivity per patient | Assessment every 12 months up to 2 years
  Dentine Hypersensitivity Experience Questionnaire: the higher the score, the greater the impact of dentin sensitivity on daily life (items have coded responses on 7-point Likert scales: 1 = "strongly disagree", 2 = "disagree", 3 = "agree a little", 4 = "neither agree nor disagree", 5 = "disagree a little", 6 = "disagree" and 7 = "strongly disagree"; a total score is then calculated)
Rate of dental surface with plaque per patient | Assessment every 3 months up to 2 years
  Recording of full mouth plaque score (FMPS) (from 0 no plaque to 100% all dental surfaces with plaque)
Rate of bleeding gingival sites per patient | Assessment every 3 months up to 2 years
  Recording of full mouth bleeding score (FMPS) (from 0 no plaque to 100% all gingival sites bleeding)

CONTACTS AND LOCATIONS:
Locations (1):
- Univeristy of Milan, Milan, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Breslin M, Taylor C. Incidence of new carious lesions and tooth loss in head and neck cancer patients: a retrospective case series from a single unit. Br Dent J. 2020 Oct;229(8):539-543. doi: 10.1038/s41415-020-2222-2. Epub 2020 Oct 23. PMID 33097891
- [Background] El-Rabbany M, Duchnay M, Raziee HR, Zych M, Tenenbaum H, Shah PS, Azarpazhooh A. Interventions for preventing osteoradionecrosis of the jaws in adults receiving head and neck radiotherapy. Cochrane Database Syst Rev. 2019 Nov 20;2019(11):CD011559. doi: 10.1002/14651858.CD011559.pub2. PMID 31745986
- [Background] Palmier NR, Migliorati CA, Prado-Ribeiro AC, de Oliveira MCQ, Vechiato Filho AJ, de Goes MF, Brandao TB, Lopes MA, Santos-Silva AR. Radiation-related caries: current diagnostic, prognostic, and management paradigms. Oral Surg Oral Med Oral Pathol Oral Radiol. 2020 Jul;130(1):52-62. doi: 10.1016/j.oooo.2020.04.003. Epub 2020 May 19. PMID 32444333
- [Background] Tao S, Zhu Y, Yuan H, Tao S, Cheng Y, Li J, He L. Efficacy of fluorides and CPP-ACP vs fluorides monotherapy on early caries lesions: A systematic review and meta-analysis. PLoS One. 2018 Apr 30;13(4):e0196660. doi: 10.1371/journal.pone.0196660. eCollection 2018. PMID 29709015